CLINICAL TRIAL: NCT03609762
Title: Effectiveness of Routine Measurement of Health-Related Quality of Life in Improving the Outcomes of Patients With Musculoskeletal Problems - A Randomized Controlled Trial
Brief Title: Effectiveness of Routine Measurement of HRQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Professor and Head of Department, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HKUCTR-2418
Record Dates: First submitted 2018-07-12; First posted 2018-08-01 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Quality of Life; Musculoskeletal Disease; Outcome
Keywords: Musculoskeletal Problems; Health-Related Quality of Life; Routine Measurement; Randomized Controlled Trial; Clinical Outcomes
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): EQ-5D-5L HRQOL results be available to the attending doctor
  Interventions: Behavioral: EQ-5D-5L HRQOL results be available to the attending doctor
- Control group (No Intervention): usual care. All subjects attending the control clinics will not need to complete the electronic EQ-5D-5L before seeing the doctor during their follow-up visits. The doctor will manage the patient as usual, based on the usual clinical information. The doctor will complete the clinician-reported follow-up clinical data form (CRF) for each subject at the end of the consultation.

INTERVENTIONS:
Behavioral: EQ-5D-5L HRQOL results be available to the attending doctor — all subjects attending the intervention clinics will complete the electronic EQ-5D-5L before seeing the doctor during each follow-up visit for the musculoskeletal problem, a print out of the longitudinal EQ-5D-5L data (Table 1) since recruitment will be given to the patients to show to the attending doctors during the consultation. The doctors will provide the management based on the usual clinical information and the additional EQ-5D-5L HRQOL results. The doctor will complete the clinician-reported follow-up clinical data form (CRF) of each eligible patient at the end of the consultation.
  Arms: Intervention group

SUMMARY:
Aim and Objectives: This is an effectiveness-implementation hybrid trial that aims to find out whether the implementation of routine measurement and reporting on the patient's EQ-5D-5L HRQOL data with an electronic platform can improve HRQOL and pain in patients with chronic knee or back problems in primary care. The investigators will also assess the acceptability of routine electronic measurement and reporting of the EQ-5D-5L in real-world primary care.

Method: This is a multi-center prospective cluster-randomized controlled trial in six public primary care clinics in Hong Kong. The six clinics will be randomized to the intervention or control group. We shall recruit 1374 (229 from each clinic) subjects with symptomatic chronic knee or back problems through the attending doctors in the clinics. Subjects of the Intervention clinics will complete the electronic EQ-5D-5L at recruitment and every follow up during the next 12 months, and a report on their longitudinal EQ-5D-5L data will be shown to the doctors during the consultations. Subjects of the control clinics will receive care as usual. All subjects will complete a set of patient reported outcome measures (PRO) including the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) on HRQOL and a 10-point Pain Rating Scale (PRS), and a structured questionnaire on sociodemographics, morbidity and service utilization rates at recruitment, and at 3, 6 and 12 months by telephone.

Outcome Measures and Data Analysis: The primary outcome is change in WOMAC total score. The secondary outcomes are change in pain, other PRO scores and doctor rated severity of disease. Group difference in changes of WOMAC and other outcome scores over time will be analyzed using generalized estimating equation model under intention-to-treat principle. The acceptability of routine measurement of HRQOL by electronic EQ-5D-5L will be analyzed by descriptive statistics.

Potential application: Routine measurement of HRQOL by an electronic EQ-5D-5L platform can be applied to other outpatient clinics to improve care of MS problems and other conditions to facilitate more effective and patient-centered care.

DETAILED DESCRIPTION:
With ageing of the population and physical inactivity in industrialized society, musculoskeletal (MS) problems have become an important disease burden, affecting hundreds of millions of people worldwide. They account for 7% of all the diagnoses presenting to primary care in Hong Kong. Although the spectrum of MS problems is broad, ranging from the common muscle strain, tendinitis and degenerative conditions to the more serious inflammatory joint diseases, they share the common characteristics of causing pain and disability. Chronic MS problems are the most common cause of severe chronic pain which impairs mental and physical well-being. The Global Burden of Disease Study 2013 (GBD 2013) showed that from 2005 to 2013, the major contributor to the global increase of disability adjusted life years (DALYs) is MS problems. Four of the top ten causes of disability in China are MS problems, namely low back pain, neck pain, osteoarthritis and other musculoskeletal problems. MS problems also significantly affect the psychosocial health of the patients' families and care givers. Current clinical management of chronic MS problems focus mainly on pain control with medications, but the outcomes are often unsatisfactory. There is increasing concern on serious side effects from the use of nonsteroidal anti-inflammatory drug (NSAID), and the risk of death and dependency from opioids in the treatment of chronic pain. More effective interventions are needed in order to reduce the suffering, disability and service burden from MS problems.

The goal of medical care is to improve or restore health. The patient's perspective need to be taken into consideration in assessing the outcome of care. Patient reported outcome (PRO) is defined as "any report of the status of a patient's health condition that comes directly from the patient, without interpretation of the patient's response by a clinician or anyone else". Pain is a commonly used PRO in clinical practice. Health-related quality of life (HRQOL) is becoming a popular PRO measure in clinical trials. HRQOL is a multidimensional concept that measures a person's subjective perceived effect on how health has affected his/her ability to live a fulfilling life, both physically and mentally. A variety of HRQOL instruments are available for different purposes, which can be generic or disease-specific. There is a large body of evidence on the psychometrics and clinimetrics of using HRQOL measures in assessing the severity of symptoms, monitoring general health and wellbeing, promoting patient-clinician communication, evaluating treatment/intervention outcomes and informing clinical decision-making. However, HRQOL is rarely measured in normal clinical practice because it requires a paradigm shift from objective to subjective outcome measures, and strategies to overcome implementation barriers of time, workload, costs and patient's burden.

The choice of instrument is critical for successful implementation of measurement of HRQOL in normal clinical practice. It should be valid, reliable, applicable to most if not all patients, short and easy to use, and meaningful. The EuroQol-5 dimension (EQ-5D) questionnaire developed by the EuroQol Group is a generic HRQOL measure that satisfies all these criteria. It consists of a descriptive system of 5 HRQOL dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a 100 mm visual analogue scale (VAS) for global health rating. It can be completed within a few minutes either by self-completion or by interview. The original EQ-5D has 3 response options to each item (EQ-5D-3L), which was modified to the EQ-5D-5L with 5 response options to each item to improve responsiveness and sensitivity9. The EQ-5D-5L has a combination of 3125 health states9. Each health state can be converted to a composite utility (preference) score from 0 (death) to 1 (perfect health), with a scoring algorithm derived from population-based valuation. The EQ-5D has been adapted to many populations with population-specific scoring algorithms available in the United States, Canada, Europe and China. A Chinese (Hong Kong) version of the EQ-5D-5L has been validated and the Hong Kong population specific EQ-5D-5L scoring algorithm has been developed from a population-based valuation study. The EQ-VAS is a 100 mm vertical scale ranging from 0 to 100, with 0 corresponding to "the worst imaginable health" and 100 indicating "the best imaginable health". Both the utility and rating scale scores are easy-to-interpret composite indicators that can be used to monitor the change in HRQOL over time. The EQ-5D-5L has been shown to be valid, reliable and sensitive in patients with MS problems internationally and in Hong Kong.

Current evidence on incorporating EQ-5D in routine clinical practice

The investigators did a systemic review from Medline and Embase databases using keywords related to HRQOL and routine clinical practice. Routine measurement of HRQOL in normal clinical practice has been used in selected patient populations, mostly in oncology and specific surgical settings in the United Kingdom (UK) and Sweden. In the UK, as a government initiative to compare service providers' performance, HRQOL has been routinely measured by the EQ-5D before and after NHS funded elective hip or knee replacement, varicose vein and inguinal hernia surgeries since 2009. This changes the paradigm of evaluation of effectiveness of care from the clinician to the patient's perspective in order to improve accountability. It also enables patients to make informed choice on service providers. In Sweden, the Swedish Hip Arthroplasty Register has recorded the EQ-5D utility score and a VAS pain score of each patient since 2002, which has demonstrated that the overall PRO of total hip replacement surgery is satisfactory, leading to a mean increase of 0.36 in EQ-5D utility score. Data on routine measurement of HRQOL by the EQ-5D or other measures in busy outpatient settings are lacking, and the investigators could not find any study on routine measurement of HRQOL in normal clinical practice in Chinese populations.

Related work done by the research team This research team has more than 20 years of experience in HRQOL research with a focus on the application of HRQOL in the evaluation of health and health services and in clinical trials. Our previous studies showed the impairment in HRQOL in people with chronic joint problems was comparable to those with chronic heart diseases and HRQOL was an important determinant of health service utilization in our Chinese population. The investigators also found that HRQOL is a responsive outcome measure of the effectiveness of interventions and quality of care in Hong Kong. Co-investigator Professor Paul Kind is one of the original authors of EQ-5D and a senior member of the EuroQoL group. He has done a lot of work on the cross-cultural adaptation of the EQ-5D and electronic administration of the EQ-5D. The investigators have developed the EQ-5D-5L utility scoring algorithm specific to the Hong Kong general population. Our pilot study on 227 Chinese patients with MS problems in a busy spine specialist outpatient clinic in Hong Kong supported the feasibility, acceptability and psychometric performance of the Chinese (Hong Kong) version of EQ-5D-5L. A limitation of our pilot study that administered the EQ-5D-5L in paper form was that the scores could not be available to the attending doctors in real-time.

In this study the investigators have developed an electronic platform for the administration, scoring and reporting of EQ-5D-5L data in normal outpatient clinics, which can make the results available to the attending doctors in real-time. The investigators have technical expertise and experience in the establishment of interactive electronic to collect PRO data with the computer or a mobile devise. The investigators have experience of using an electronic platform for the administration of questionnaire and collection of both patient reported and clinical data from multiple study sites in a health services project for low income families. Our team has also developed an interactive Mobile App to promote exercise and to collect data on usage.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 18 years or above
2. b) has doctor-diagnosed symptomatic knee and/or back pain problem that is expected to last for one month or more
3. scheduled for at least one follow-up visits in the clinic within 12 months
4. has given written consent to participate in this study

Exclusion Criteria:

1. life expectancy less than 12 months (judged by the doctor),
2. has cancer
3. too ill (both physically or cognitively) to complete a questionnaire
4. unable to communicate in Chinese
5. does not give consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1374 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The change in HRQOL measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) global score | At baseline, and 3 months, 6 months and 12 months after baseline
  The WOMAC is a widely used condition specific HRQOL measure to assess pain, stiffness and physical function of patients with MS problems. It has been applied to patients with hip and/or knee osteoarthritis, low back pain, rheumatoid arthritis and fibromyalgia. It consists of 24 items on 3 domains: pain (5 items), stiffness (2 items) and physical function (17 items). Each question is rated on a 5-point Likert scale from 0 to 4, with lower scores indicating lower levels of symptoms or impairment. The item scores in each domain subscale are summated to a domain score. The global WOMAC score is calculated by summating the three domain scores. A Chinese version of WOMAC is available and has been shown to be valid, reliable and sensitive in Chinese patients.

SECONDARY OUTCOMES:
The change in pain score measured by the 10-point Pain Scale | At baseline, and 3 months, 6 months and 12 months after baseline
  The patient will be asked to rate their pain that best represents the intensity of their pain using a scale from 0 to 10, where 0 indicates no pain and 10 indicates the worse pain.
The change in patient-reported outcomes (PRO) - SF-6D utility score | At baseline, and 3 months, 6 months and 12 months after baseline
  The SF-6D is a preference-based measure of health, derived from the SF-36 Health Survey, that generates a utility score. It has 6 items measuring six HRQOL dimensions of physical function (PF), role limitation (RL), social functioning (SF), bodily pain (BP), mental health (MH) and vitality (VT). The SF-6D responses have a combination of 18,000 health states. Each health state can be converted to a composite preference (utility) score from 0 indicating death to 1 indicating perfect health. The Chinese SF-6D was validated in the Chinese population in Hong Kong, and the Hong Kong population-based scoring algorithm was established. The mean SF-6D utility score of the Hong Kong Chinese population is 0.78.
The change in patient-reported outcomes (PRO) - global health measured by the Global Rating Scale (GRS) | At baseline, and 3 months, 6 months and 12 months after baseline
  The GRS on change in health will be used to assess the patient's self-perception of any change in the overall health condition on a 7-point scale: (-3,(much worse), -2 (worse), -1 (a little worse), 0 (no change), 1 (a little better), 2 (better), and 3 (much better)).
The change in patient-reported outcomes (PRO) - patient enablement measured by the Patient Enablement Instrument (PEI) score | At baseline, and 3 months, 6 months and 12 months after baseline
  The PEI is a 6-item questionnaire that measures the patient's perceived change in coping with illness and self-care. Each item is rated on a 3-point (0, 1, and 2) scale. The sum of the item scores gives the final PEI score, with higher scores indicating better enablement. The Chinese version was shown to be a valid, reliable and sensitive outcome measure among Chinese patients in Hong Kong.
The change in clinician-reported disease severity | At baseline, and 3 months, 6 months and 12 months after baseline
  The diagnosis and duration of the chief musculoskeletal problem will be reported by the attending doctor. The attending doctor will rate patient's disease severity on a 5-point Likert scale: 1. no problem, 2. mild, 3. moderate, 4. severe and 5.very severe.
The change in clinician-reported disease progression | At baseline, and 3 months, 6 months and 12 months after baseline
  The diagnosis and duration of the chief musculoskeletal problem will be reported by the attending doctor. In each follow-up clinic consultation, the attending doctor will rate patient's disease progression on a 7-point scale (-3 much worse, -2 worse, -1 a little worse, 0 no change, 1 a little better, 2 better, and 3 much better).

OTHER OUTCOMES:
Difference in the health service utilization rates between intervention group and control group | At baseline, and 3 months, 6 months and 12 months after baseline
  Health service utilization included monthly frequency of outpatient consultations with western/Chinese medicine practitioners, allied health service visits, accident and emergency (A&E) department attendance, and admissions to hospitals.
Difference in the drug and other treatment utilization rates between intervention group and control group | At baseline, and 3 months, 6 months and 12 months after baseline
  Medication use in the past one month will be asked in the survey to evaluate the drug treatment utilization rates.
Difference in the patient acceptability of routine measurement of HRQOL by the electronic EQ-5D-5L between intervention group and control group | At baseline, and 3 months, 6 months and 12 months after baseline
  The acceptability of routine completion of the electronic EQ-5D-5L will be evaluated by the perceived ease of use and perceived usefulness scales based on the Technology Acceptability Model (TAM), which was translated and validated on the local Chinese population.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L. K. LAM, Principal Investigator — Professor and Head
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
On completion of the trial, and after publication of the primary manuscript, data requests can be submitted to corresponding author at The Department of Family Medicine and Primary Care, The University of Hong Kong.
Time Frame: On completion of the trial, and after publication of the primary manuscript
Access Criteria: Will be assessed by the corresponding author at The Department of Family Medicine and Primary Care, The University of Hong Kong

REFERENCES:
- [Derived] Ng APP, Liu KSN, Cheng WHG, Wong CKH, Cheng JKY, Lam JSM, Or CK, Tse ETY, Lam CLK. Feasibility and acceptability of electronic EQ-5D-5L for routine measurement of HRQOL in patients with chronic musculoskeletal problems in Hong Kong primary care. Health Qual Life Outcomes. 2022 Sep 20;20(1):137. doi: 10.1186/s12955-022-02047-0. PMID 36127713
- [Derived] Lam C, Chin WY, Wong CKH, Or K, Fong DYT, Cheung JPY, Chao DVK, Wong ELY, Kind P. Effectiveness of routine measurement of health-related quality of life in improving the outcomes of patients with musculoskeletal problems-a cluster randomised controlled trial: protocol paper. BMJ Open. 2020 Dec 15;10(12):e040373. doi: 10.1136/bmjopen-2020-040373. PMID 33323434
- See also: protocol paper — http://bmjopen.bmj.com/cgi/content/full/bmjopen-2020-040373
- See also: electronic EQ-5D-5L psychometrics — https://doi.org/10.1186/s12955-021-01898-3
- See also: Feasibility & acceptability of electronic EQ-5D-5L — https://doi.org/10.1186/s12955-022-02047-0
- See also: Enablement mediates between pain and HRQOL — https://doi.org/10.3399/BJGP.2022.0546